CLINICAL TRIAL: NCT01366157
Title: Investigation to Evaluate the Levels of Human Germinal-center-Associated Lymphoma (HGAL) Protein in Pediatric Hodgkin Lymphoma and Correlate With Early Response
Brief Title: Protein Biomarker Levels in Tissue Samples From Young Patients With Low-risk Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AHOD11B1; COG-AHOD11B1 (Other: Children's Oncology Group); CDR0000701020 (Other: Clinical Trials.gov); NCI-2011-02859 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Lymphoma
Keywords: childhood favorable prognosis Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; childhood lymphocyte depletion Hodgkin lymphoma; childhood lymphocyte predominant Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma; childhood nodular lymphocyte predominant Hodgkin lymphoma; childhood nodular sclerosis Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research trial is studying protein biomarker levels in tissue samples from young patients with low-risk Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the variability of expression of human geminal-center-associated lymphoma (HGAL) protein in pediatric low-risk Hodgkin lymphoma.
* To assess the variability of HGAL staining between risk groups by comparing samples from subjects enrolled in the low-risk study AHOD0431 with subject samples enrolled in AHOD0031 for intermediate-risk classical Hodgkin Lymphoma (cHL).
* To assess the variability of HGAL staining by evaluating a tissue array created from subjects with intermediate-risk cHL.
* To correlate rapid or slow early-response in the intermediate-risk group with HGAL protein expression.

OUTLINE: Paraffin-embedded tissue samples and tissue microarrays are analyzed for protein expression by IHC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with low-risk classical Hodgkin lymphoma (cHL)
* Samples available from patients enrolled in the low-risk study COG-AHOD0431 and in the intermediate-risk cHL study COG-AHOD0031

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosed with low-risk classical Hodgkin lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Variability of HGAL protein expression in pediatric patients with low-risk classical Hodgkin lymphoma (cHL)
Variability of HGAL staining between low-risk and intermediate-risk pediatric patients with cHL
Variability of HGAL staining as assessed by tissue array in pediatric patients with intermediate-risk cHL
Correlation of rapid or slow early response in the intermediate-risk group with HGAL protein expression

CONTACTS AND LOCATIONS:
Overall Officials: Frank G. Keller, MD, Principal Investigator — Emory Children's Center - Atlanta